CLINICAL TRIAL: NCT00176605
Title: A Phase II Trial of Metronomic Dosing of Etoposide and Cyclophosphamide in Patients With Stage D0 Prostate Cancer.
Brief Title: Phase II Metronomic Dosing, Etoposide, Cyclophosphamide, D0 Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080408; P30CA072720 (NIH); 0220044931 (Other: IRB Number); CDR0000443482; NCT00227643 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Etoposide; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Etoposide + Cyclophosphamide) (Experimental): Therapy will be divided into 4 cycles. Each cycle will be composed of 6 weeks of therapy. Total duration of therapy is 24 weeks. Administration of etoposide (50 mg po qd) and cyclophosphamide (50 mg po qd) will alternate in 21 day intervals. Starting with etoposide, patients will receive 21 days of therapy, upon completion of etoposide therapy patients will then receive 21 days of cyclophosphamide therapy. Therapy will continue in this alternating manner for 24 weeks. Week 1 of each cycle, begins with etoposide; Week 4 of each cycle, begins with cyclophosphamide.
  Interventions: Drug: Etoposide; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Etoposide — 50 mg per day of Etoposide orally for 21 consecutive days. Etoposide will be alternated with oral cyclophosphamide. The drug is administered at night just prior to bed. Week 1 of each cycle will begin with etoposide.
Drug: Cyclophosphamide — 50 mg per day of cyclophosphamide orally for 21 consecutive days. Cyclophosphamide will be alternated with oral etoposide. The drug is taken 2 hours after breakfast. The patient will be asked to increase hydration throughout the day. Recommendation is at least 6, 8oz glasses of water or other non-caffeinated beverage. Week 4 of the each cycle will begin with cylcophosphamide. Chronic administration of cyclophosphamide at this dose has been well tolerated

SUMMARY:
Based on data supporting the use of cyclophosphamide and etoposide both as single agents in combination and a Phase I study showing acceptable toxicity with a chronic dosing regimen, we propose a Phase II clinical trial. This protocol establishes a model that will test the hypothesis that the use of etoposide and cyclophosphamide early in the course of prostate cancer progression, when fewer tumor cells are present, will have greater anti-tumor activity. We plan to treat patients with stage D0 prostate cancer to assess toxicity and anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria

* Patients with histologically proven prostate cancer and tumors limited to the prostate (including seminal vesicle involvement, provided all visible disease was surgically removed) that have completed local therapy and have an rising PSA value, as defined in Section 5.1.5.
* Prior androgen ablation therapy is allowed as long as the patient completed therapy at least 1 year prior to entry into this study. The patient must be fully recovered from such therapy and must not have demonstrated progression while on androgen ablation therapy.
* Primary treatment to the prostate (surgery and/or radiation) must have been completed at least 3 months prior to entry into this study and the patient must be fully recovered from such therapy.
* Patients must have a negative CT of the chest, abdomen and pelvis and bone scan. The scans must be completed within 4 weeks prior to the date of starting therapy.
* PSA value for patients enrolled must be > 2 ng/ml with a doubling time of £ 12 months. PSA value > 2 ng/ml must be documented by two measurements at least four weeks apart. The final PSA measurement before study entry must be obtained within one week prior to therapy. This will be considered the baseline PSA. (Note: The website http://www.mskcc.org/mskcc/html/10088.cfm may be used to access a prostate normogram calculator.)
* The following lab values must be obtained within 4 weeks prior to therapy:
* ANC ≥1500/mm³,
* Hemoglobin ≥ 10 g/dl
* Platelet count ≥ 100,000/mm³
* Serum creatinine ≤ 1.5 mg/dL
* Total bilirubin ≤ 1.5 mg/dL
* Liver function tests (SGOT, SGPT) ≤ 1.5 times the upper limit of the institution's normal range.
* Men ≥ 18 years of age.
* An estimated life expectancy of at least 6 months.
* ECOG performance status ≤ 2.
* Able to give informed, written consent.
* Men must consent to using effective contraception (barrier method- latex condom) while on treatment and for 4 weeks after discontinuation of treatment.

Exclusion Criteria

* Patients with active infections or known infection with HIV (HIV testing will not be performed as part of this study).
* Any coexisting medical condition including uncontrolled cardiac, hepatic, renal or psychiatric disease defined as ³ Grade 3 (CTCAE Version 3).
* Concurrent use of other investigational agent.
* Patients that have previously received more than 2 months of therapy with any of the agents used in this study.
* PSA value < 2 ng/ml.
* Prior chemotherapy in the past 5 years.
* Use of androgen ablation therapy within 1 year, or history of progression on androgen ablation therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stein, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (7):
- United States (7):
  - Central Jersey Oncology Center, East Brunswick, New Jersey
  - Robert Wood Johnson University Hospital/CINJ at Hamilton, Hamilton, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - UMDNJ/Robert Wood Johnson Medical School, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Cancer Institute of New Jersey (a comprehensive cancer center at an academic institution) and Robert Wood Johnson University Hospital at Hamilton (a community hospital) from August 2005 through May 2008.
Groups:
- Arm 1 (Etoposide + Cyclophosphamide): Therapy will be divided into 4 cycles. Each cycle will be composed of 6 weeks of therapy for a total of 24 weeks. Administration of etoposide (50 mg po qd) and cyclophosphamide (50 mg po qd) will alternate in 21 day intervals. Starting with etoposide, patients will receive 21 days of therapy, upon completion of etoposide therapy patients will then receive 21 days of cyclophosphamide therapy. Week 1 of each cycle, begins with etoposide; Week 4 of each cycle, begins with cyclophosphamide.
  Cyclophosphamide : 50 mg per day of cyclophosphamide orally for 21 consecutive days. Cyclophosphamide will be alternated with oral etoposide. The drug is taken 2 hours after breakfast. The patient will be asked to increase hydration throughout the day. Recommendation is at least 6, 8oz glasses of water or other non-caffeinated beverage. Week 4 of the each cycle will begin with cylcophosphamide. Chronic administration
Period: Overall Study
Arm/Group | Arm 1 (Etoposide + Cyclophosphamide)
Started | 15
Completed | 13
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1 (Etoposide + Cyclophosphamide)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: PSA Response Rate
Description: The PSA response rate is the percentage of patients who have a PSA response. A PSA response will be considered a PSA decline of at least 50% must be confirmed by a second PSA value four or more weeks later. The reference PSA for these declines should be a PSA measured within 2 weeks prior to the initiation of therapy. Patients may not demonstrate clinical or radiographic evidence of disease progression during this period.
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 (Etoposide + Cyclophosphamide)
Number analyzed (Participants) | 13
percentage of participants | 15.4

2. Secondary Outcome: Toxicities Related to Chronic Administration of Etoposide and Cyclophosphamide in Patients With Stage D0 Prostate Cancer.
Description: All patients who receive one dose of protocol therapy will be evaluable for toxicity. A total of 15 patients received at least one dose of protocol therapy. Adverse events are described in Adverse Event section.
Time Frame: 5 years
Population: No subjects experienced serious adverse events related to the intervention.
Measure: Number; unit: participants
Arm/Group | Arm 1 (Etoposide + Cyclophosphamide)
Number analyzed (Participants) | 15
participants | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Arm 1 (Etoposide + Cyclophosphamide)
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Etoposide + Cyclophosphamide) (N=15)
Valvular heart disease (Cardiac disorders) | 1 (1) — Patient admitted for sycopy. Cardiac workup showed critical aortic valve stenosis. Unlikely related to protocol.
Ulcer, GI - Anus (Gastrointestinal disorders) | 1 (1) — Perirectal abscess
Infection with unknown ANC - appendix (Infections and infestations) | 1 (1) — Unlikely related to protocol.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Etoposide + Cyclophosphamide) (N=15)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (4)
Anorexia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (astenia, lethary, malaise) (General disorders) | 6 (6)
Constitution Symptoms (Other) (General disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (1)
Sweating (diaphoresis) (General disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Pain/ - head/headache (General disorders) | 4 (4)
Pain - chest/thorax NOS (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Mood alteration - depression (Psychiatric disorders) | 1 (2)
Neuropathy: sensor (Nervous system disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes